CLINICAL TRIAL: NCT00486317
Title: SMC021A - Absorption, Efficacy and Tolerance in Patients With Osteoarthritis. A Placebo-Controlled 14-Days Study.
Brief Title: Pharmacokinetics/Pharmacodynamics of Oral Salmon Calcitonin in Patients With Osteoarthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nordic Bioscience A/S (Industry)
Collaborators: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMC021A2110
Record Dates: First submitted 2007-06-13; First posted 2007-06-14 (Estimated); Last update posted 2007-06-14 (Estimated); Status verified 2007-06

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis, oral salmon calcitonin, tolerability, biomarkers
MeSH Terms: conditions — Osteoarthritis | interventions — salmon calcitonin

INTERVENTIONS:
Drug: Oral salmon calcitonin, salmon calcitonin nasal spray

SUMMARY:
The purpose of this study is to expose patients with OA to calcitonin and to determine plasma calcitonin levels after administration of 0.6 mg and 0.8 mg oral calcitonin and 200 IU nasal calcitonin. Also the purpose is to assess the effect of different doses of oral calcitonin (0.6 mg and 0.8 mg oral) and 200 IU nasal calcitonin compared to placebo on serum CTX-I and CTX-II. Finally to assess the tolerance profile of different doses/formulations of oral calcitonin compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Medical history and symptoms of knee osteoarthritis

Exclusion Criteria:

* Any other disease or medication affecting the bone or cartilage.
* Any clinical signs or laboratory evidence diseases, which in the Investigator's opinion would preclude the participant from adhering to the Protocol or completing the trial.

Ages: 52 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2005-10

PRIMARY OUTCOMES:
Number of adverse events

SECONDARY OUTCOMES:
Changes in Urine CTX-I and CTX-II
Changes in serum osteocalcin

CONTACTS AND LOCATIONS:
Overall Officials: Bente J Riis, M.D., Study Chair — Nordic Bioscience A/S
Locations (1):
- CCBR A/S, Ballerup Municipality, Denmark